CLINICAL TRIAL: NCT00062322
Title: Phase I Study of Preoperative Chemo/Radiation (Concurrent Irinotecan/Cisplatin/RT) Followed by Surgery in Limited Stage Small Cell Lung Cancer (SCLC-LS)
Brief Title: Neoadjuvant Chemoradiotherapy Followed By Surgery in Treating Patients With Limited-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000304720; P30CA006927 (NIH); FCCC-02613
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Irinotecan; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: irinotecan hydrochloride
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as irinotecan and cisplatin use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Irinotecan and cisplatin may also make the tumor cells more sensitive to radiation therapy. Combining chemotherapy with radiation therapy before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: This phase I trial is studying the side effects of neoadjuvant radiation therapy given together with irinotecan and cisplatin followed by surgery in treating patients with limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and feasibility of neoadjuvant chemoradiotherapy with irinotecan and cisplatin followed by surgery in patients with limited stage small cell lung cancer.
* Determine the pathologic complete response rate of patients treated with this regimen.
* Correlate the level of vascular endothelial growth factor with treatment response and disease outcome in patients treated with this regimen.
* Correlate genetic polymorphisms in cytochrome P450 1A1, glutathione S-transferase M1 and P1, myeloperoxidase, and NAD(p)H: quinone oxidoreductase with treatment response and disease outcome in patients treated with this regimen.

OUTLINE: This is a pilot study.

* Induction chemotherapy: Patients receive cisplatin IV over 1 hour on day 1 and irinotecan IV over 90 minutes on days 1 and 8.
* Chemoradiotherapy: Beginning on day 21, patients receive chemoradiotherapy comprising radiotherapy once daily, 5 days a week for 4 weeks and then twice daily for 4 days. Patients also receive cisplatin IV and irinotecan IV over 30-60 minutes once weekly concurrently with radiotherapy. Treatment continues in the absence of disease progression or unacceptable toxicity.

At the completion of chemoradiotherapy, patients are evaluated for surgery. Patients who are candidates for surgery receive one additional course of cisplatin IV and irinotecan IV. Patients who are not candidates for surgery receive radiotherapy twice daily for 4 days and cisplatin IV and irinotecan IV as in chemoradiotherapy.

* Surgery: Approximately 2-4 weeks after the last dose of chemotherapy, patients undergo surgery.

Patients are followed every 4 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer

  * Limited stage disease (clinical stage I-IIIA) and meets the following criteria:

    * Confined to 1 hemithorax
    * No T4 disease based on malignant pleural effusion
    * No N3 disease based on contralateral hilar or supraclavicular involvement
  * Contralateral mediastinal (N3) nodes greater than 1.5 cm on CT scan must be biopsied to rule out pathologic involvement
* Measurable or evaluable disease
* Tumor must be able to be encompassed by limited radiotherapy field without significantly compromising pulmonary function
* No pleural effusion visible on chest x-ray (regardless of cytology)
* No prior complete tumor resection

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count at least 1,800/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* No known Gilbert's disease

Renal

* Creatinine no greater than 1.5 mg/dL
* Calcium less than 12.0 mg/dL

Cardiovascular

* No myocardial infarction within the past 6 months
* No congestive heart failure
* No uncontrolled arrhythmias
* No active unstable angina

Pulmonary

* Calculated postoperative FEV_1 at least 800 cc
* No chronic obstructive pulmonary disease with FEV_1 no greater than 1 L or uncontrolled bronchospasm in the unaffected lung

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 2 years except curatively treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or any other noninvasive malignancy
* No history of seizures
* No history of uncontrolled psychiatric illness that would preclude giving informed consent or complying with study
* No active or uncontrolled infection
* No uncontrolled diabetes mellitus (random blood sugar at least 250 mg/dL)
* No other concurrent serious medical illness
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior irinotecan
* No prior topotecan

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the chest or other areas containing 30% or more of marrow-bearing bone

Surgery

* See Disease Characteristics

Other

* No concurrent phenytoin, phenobarbital, or other antiepileptic prophylactic drugs
* No concurrent amifostine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-02; Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Feigenberg, MD, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States